CLINICAL TRIAL: NCT02929706
Title: Effectiveness of Thiopurine Dose Optimization by NUDT 15 R139C on Reducing Thiopurine-induced Leucopenia in Inflammatory Bowel Disease
Brief Title: Pre-genotype NUDT 15 R139C on Reducing Thiopurine-induced Leucopenia in Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20160704
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2016-10

CONDITIONS: Thiopurine-induced Leukopenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- intervention group (Experimental): Pre-genotype NUDT15 and optimize azathioprine dosage.The wild type use azathioprine(Imuran，2-2.5mg/kg/d),the CT genotype use half dose of azathioprine（Imuran，1-1.5mg/kg/d).The TT genotype avoid use of azathioprine.
  Interventions: Genetic: Pre-genotype NUDT15 and optimize azathioprine dosage
- control group (No Intervention): optimize the thiopurine use by coventional strategy without konwing NUDT15 genotype

INTERVENTIONS:
Genetic: Pre-genotype NUDT15 and optimize azathioprine dosage — Pre-genotype NUDT15 and optimize azathioprine dosage.The wild type use azathioprine(Imuran，2-2.5mg/kg/d),the CT genotype use half dose of azathioprine（Imuran，1-1.5mg/kg/d).The TT genotype avoid use of azathioprine.
  Arms: intervention group

SUMMARY:
NUDT15 R139C was comfirmed to be associated with thiopurine-induced leukopenia inflammatory bowel disease (IBD) cohort.The present study aim to explor the following questions:can optimizing thiopurine dose by NUDT15 genotype reduce thiopurine-induced leucopenia?What is the influence of this optimizing strategy on clinical outcome?Thus,we conduct a randomised controlled study.Subject in the conventional group detect NUDT15 genotype before thiopurine use and optimise dosage according to the genotype.While the subjects in the control group follow the conventional monitor strategy.The primary endpoint was the rate of leukopenia.The secondary endopoint was the efficacy of thiopurine.The follow up duration was 1 year.

DETAILED DESCRIPTION:
We included patients diagnosis of IBD (>18 yrs old) with indication of the use of thiopurine.Group A (intervention): AZA dose optimization by testing for NUDT15 R139C- testing results will be informed.Group B (control):AZA dose optimization according to standard guideline - testing results will not be informed.The participants will be followed for 9 month. The incidence of adverse events and efficacy will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IBD with indication of the use of thiopurine

Exclusion Criteria:

* Contraindication of thiopurine
* Previous use of thiopurine
* co-treatment with 5-ASA or allopurinol

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
difference of incidence of leucopenia ADR | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523
- [Derived] Chao K, Huang Y, Zhu X, Tang J, Wang X, Lin L, Guo H, Zhang C, Li M, Yang Q, Huang J, Ye L, Hu P, Huang M, Cao Q, Gao X. Randomised clinical trial: dose optimising strategy by NUDT15 genotyping reduces leucopenia during thiopurine treatment of Crohn's disease. Aliment Pharmacol Ther. 2021 Nov;54(9):1124-1133. doi: 10.1111/apt.16600. Epub 2021 Sep 25. PMID 34563096